CLINICAL TRIAL: NCT04443309
Title: A Single-arm, Non-randomized, Single-center Study to Evaluate Lenvatinib in Combination With Camrelizumab as First-Line Therapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Lenvatinib in Combination With Camrelizumab as First-Line Therapy in Patients With Advanced HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2286
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib plus Camrelizumab (Experimental): Camrelizumab (Jiangsu HengRui Medicine Co., Ltd.) is a recombinant anti-human PD-1 IgG4 monoclonal antibody.
  Lenvatinib is a novel angiogenesis inhibitor which targets multiple tyrosine kinases， including vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT.
  Interventions: Drug: Camrelizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg,iv,d1,q2w
  Other Names: SHR-1210
Drug: Lenvatinib — Lenvatinib 8mg (<60kg) or 12mg (≥60kg),po,d2,qd
  Other Names: LENVIMA,E7080

SUMMARY:
This is a single arm, open-label, non-randomized and single-center phase I/II clinical study, to evaluate the the safety, tolerance and efficacy of Lenvatinib plus Camrelizumab as first-line therapy in patients with advanced Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerance and efficacy of Lenvatinib combined with Camrelizumab as first-line therapy for patients with advanced hepatocellular carcinoma.The target sample size is 53.In the first phase 6 panticipants was evaluated (N=3+3), If there was no obvious dose-limiting toxicity (DLT), then entered the extended phase (N=47).Treatment continually until disease progression or intolerable toxicity or patients withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol;
2. Males or females, age ≥ 18 years at the time of informed consent;
3. Imaging (by AASLD or Standard for the diagnosis and treatment of primary liver cancer 2017 in China) or histopathologically or cytologically confirmed advanced HCC;
4. BCLC stage B or C, and not suitable for surgical or local therapy, or has progressed following surgical and/or local therapy;
5. No previous systematic treatment for HCC;
6. Have at least one measurable lesion (in accordance with RECIST v1.1); the measurable lesion has a long diameter ≥ 10 mm or lymphadenopathy has a short diameter ≥ 15 mm in spiral CT scan;
7. ECOG-PS score 0 or 1
8. Child-Pugh Class: Grade A
9. Life Expectancy of at least 3 months
10. Subjects with HBV infection: HBV DNA<2000 IU/ml or <10^4 copy/mL, and have received anti-HBV therapy for at least 14 days prior to enrollment in the study, subjects with HCV-RNA(+) must receive antiviral therapy;
11. Hematology and organ functions are sufficient based on the following laboratory results within 14 days prior to the treatment of this study:

    Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): WBC ≥ 3.0×10^9/L, HB ≥ 85 g/L; Neutrophils ≥ 1.5×10^9/L; PLT≥75×10^9/L; Biochemical examination (no ALB infused within 14 days): ALB ≥ 29 g/L; ALP and ALT and AST < 5×ULN; TBIL≤3×ULN; Adequate renal function: Cr≤1.5×ULN, or CCr>50mL/min; Female: CrCl = ((140- year) x weight (kg) x 0.85)/72x Cr (mg/dL) Male: CrCl = ((140- year) x weight (kg) x 1.00)/72xCr (mg/dL)
12. Agree to abstain from sex (avoid heterosexual intercourse) or use contraceptive methods with an annual contraceptive failure rate of less than 1% during treatment and for at least 6 months after the last administration.

Exclusion Criteria:

1. Hepatocellular carcinoma patients with any of the following:

   Suitable for radical surgery; without an assessment lesion after radical surgery; liver transplantation history or ready for liver transplantation;
2. History of hepatic encephalopathy;
3. Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma;
4. Pregnant women (positive pregnancy test before taking medicine) or lactating women;
5. Known history of serious allergy to any monoclonal antibody or targeted anti-angiogenic drug (or any excipient);
6. Received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection;
7. Previous or existing CTCAE 5.0 standard grade 3 or above gastrointestinal fistula or non-gastrointestinal fistula (such as skin);
8. Factors to affect oral administration and absorption (such as inability to swallow, chronic diarrhea and intestinal obstruction);
9. Ascites with clinical symptoms (i.e. ascites with Child-Pugh rating > 2) or cancerous ascites require therapeutic abdominal puncture or drainage. Or uncontrolled malignant ascites (ascites that researchers believe diuretics or puncture cannot control);
10. Major surgical operations (except biopsy) were performed within 4 weeks prior to the first study of drug therapy or the surgical incision was not completely healed; Minor surgery (i.e. simple resection, biopsy, etc.) was performed within 7 days before the first round of research intervention.
11. Cardiovascular and cerebrovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accident or transient ischemic attack, congestive heart failure occurred within 6 months prior to admission (New York Heart Association Grade ≥2, see Appendix 4); Arrhythmia requiring antiarrhythmic drugs (except β receptor blocker or digoxin); Repeated ECG detection QTcF interval>480 milliseconds (ms).
12. Hepatic and renal insufficiency, such as jaundice, ascites, and/or bilirubin>3×ULN, creatinine ratio>3.5g/24h, or renal failure requiring blood or peritoneal dialysis, etc. And/or urine routine showed proteinuria ≥++or confirmed 24-hour proteinuria>1.0g.
13. Persistent>2 grade (CTC-AE5.0) infection.
14. History of thromboembolism (including stroke and/or transient ischemic attack) in the past 6 months.
15. Hypertension (systolic blood pressure>160mmHg, diastolic blood pressure>100 mmHg) that not be well controlled through antihypertensive drug treatment.
16. History of active autoimmune diseases or autoimmune diseases in the past two years.
17. Known central nervous system metastasis and/or cancerous meningitis.
18. Be ready for or previously received organ or allogenic bone marrow transplantation.
19. Known history of active tuberculosis (Mycobacterium tuberculosis).
20. History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage.
21. History of human immunodeficiency virus (HIV)infection.
22. Active hepatitis B virus or C virus infection and not receive regular treatment;
23. Serious non-healing wound, ulcer or fracture.
24. Drug abuse exists; or any medical, psychological or social condition that may affect research, unstable patient compliance or even endanger patient safety.
25. Any>1 grade (CTC-AE 5.0) unresolved toxicity due to previous treatment or operation, except for hair loss, anemia, and hypothyroidism.
26. Previous and current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and severe impairment of lung function.
27. Received a potent CYP3A4 inhibitor treatment within 7 days prior to the study or received a potent CYP3A4 inducer within 12 days prior to the study.
28. With other active malignant tumors except HCC within 5 years or simultaneously.
29. Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.
30. Patients participate in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | one year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | one year
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit
Progression-free Survival (PFS) | one year
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause
Overall Survival (OS) | one year
  Duration from the date of initial treatment to the date of death due to any cause.
Duration of Response (DOR) | one year
  Duration from the first time reported partial response or complete response to the first time of disease progression or death
Clinical Benefit Rate (CBR) | two years
  Proportion of patients achieved complete response and partial response for more than 6 months
3-months and 6-months Progression Free Survival Rate | 6 months
  Portion of patients who do not experience disease progression (defined by RECIST 1.1) or death of any cause after treated with toripalimab plus lenvatinib for 3 months and 6 months
6-months and 1-year Mortality Rate | one year
  Portion of patients who die of any cause after treated with toripalimab plus lenvatinib at 6 months and 1 year, respectively
Adverse Events (AE) | two years
  Any adverse events related with treatment drugs and details include adverse events type, frequency and severity

OTHER OUTCOMES:
Biomarker | two years
  Biomarkers (such as AFP, PD-L1 expression, CD8 T cell immunohistochemistry, RNA-sequencing) related with efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Please Select, China

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Llovet JM, Montal R, Villanueva A. Randomized trials and endpoints in advanced HCC: Role of PFS as a surrogate of survival. J Hepatol. 2019 Jun;70(6):1262-1277. doi: 10.1016/j.jhep.2019.01.028. Epub 2019 Mar 31. PMID 30943423
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] 8. Qin S OX, Bai Y, Cheng Y, Chen Z, Ren Z, Song T, Dutcus C, Saito K, Tamai T, Yau TCC, Rau K-M, Cheng A-L, Han G. Subgroup analysis of Chinese patients in a phase 3 study of lenvatinib vs sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma. Hepatol Int 2019;13:S170.
- [Background] Boussiotis VA. Molecular and Biochemical Aspects of the PD-1 Checkpoint Pathway. N Engl J Med. 2016 Nov 3;375(18):1767-1778. doi: 10.1056/NEJMra1514296. No abstract available. PMID 27806234
- [Background] Ma W, Gilligan BM, Yuan J, Li T. Current status and perspectives in translational biomarker research for PD-1/PD-L1 immune checkpoint blockade therapy. J Hematol Oncol. 2016 May 27;9(1):47. doi: 10.1186/s13045-016-0277-y. PMID 27234522
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738